CLINICAL TRIAL: NCT06011876
Title: Genetic Biomarkers of Intermittent Hypoxia-Induced Respiratory Motor Plasticity in Chronic SCI
Brief Title: BioFLO for Respiratory Recovery in SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202202891; W81XWH2210478 (Other Grant/Funding Number: US ARMY MED RES ACQUISITION)
Record Dates: First submitted 2023-08-01; First posted 2023-08-25 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries
Keywords: acute intermittent hypoxia; spinal cord injury; breathing; motor function
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-session testing days (Experimental): Participants will complete three separate single-session testing days. Baseline testing will be performed, then on each day, participants will receive AIH, AIHH, and sham AIH in random order. Post-testing will occur after each intervention.
  Interventions: Other: Acute Intermittent Hypoxia (AIH); Other: Acute Intermittent Hypercapnic-Hypoxia (AIHH); Other: Sham AIH
- Respiratory strength training blocks (Experimental): Participants will complete three separate respiratory strength training blocks. In each block, participants will receive 5 days of AIH, 5 days of AIHH, and 5 days of sham AIH in random order, followed by respiratory strength training. Each block will include 5 days of intervention and training, and post-testing 1, 3, and 7 days after intervention and training has concluded.
  Interventions: Other: Acute Intermittent Hypoxia (AIH); Other: Acute Intermittent Hypercapnic-Hypoxia (AIHH); Other: Sham AIH

INTERVENTIONS:
Other: Acute Intermittent Hypoxia (AIH) — AIH (acute intermittent hypoxia) consists of short episodes of low oxygen (9% O2).
Other: Acute Intermittent Hypercapnic-Hypoxia (AIHH) — AIHH consists of short episodes of low oxygen (9% O2) and elevated carbon dioxide (4% CO2).
Other: Sham AIH — A single session of sham AIH with episodes of normal room air (21% O2).

SUMMARY:
Acute intermittent hypoxia (AIH) involves brief (1 min), repeated episodes (~15) of breathing low oxygen air to stimulate spinal neuroplasticity. Animal and human studies show that AIH improves motor function after spinal cord injury, particularly with slightly increased carbon dioxide (hypercapnic AIH; AIHH) and task-specific training. Using a double blind cross-over design, the study will test whether AIHH improves breathing more than AIH and whether specific genetic variations are related to individuals' intervention responses.

DETAILED DESCRIPTION:
This study will consist of two parts - single-session testing days, and respiratory strength training blocks. If a participant is not eligible to enroll in single-day testing, they will be asked to enroll in only the respiratory strength training blocks.

On single-session testing days, participants will be asked to come in on three separate days they will complete a battery of tests, then be given one of three interventions, and then complete the same battery of tests. The three interventions are acute intermittent hypoxia (AIH), acute intermittent hypercapnic-hypoxia (AIHH), or sham acute intermittent hypoxia (sham AIH). These interventions are explained in more detail below.

During respiratory strength training blocks, participants will receive five days of AIH, AIHH, or sham AIH in combination with respiratory strength training, which uses small hand-held devices to strengthen the muscles used for breathing. Participants will be asked to complete all three blocks to receive all three interventions. In addition to 5 days of interventions and respiratory strength training, the respiratory strength training blocks include testing 1 day, 3 days, and 7 days after the 5 days of respiratory strength training.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18-70 years of age
2. Chronic incomplete SCI ≥ 1 year at or below C1-T12

   * Incomplete SCI based on residual sensory and motor function below the level of the injury or injury classification of B, C, D at initial screening according to the American Spinal Injury Association Impairment Classification and the International Standards for the Neurological Classification of SCI.

   -OR- Chronic complete SCI ≥1 year at or below C4-T12
   * Complete SCI based on the absence of residual sensory or motor function below the level of injury or injury classification of A at initial screening according to the American Spinal Injury Association Impairment Classification and the International Standards for the Neurological Classification of SCI.
3. Medically stable with physician clearance
4. SCI due to non-progressive etiology
5. 20% impairment in maximal inspiratory, maximal expiratory pressure generation, or both relative to normative values

Exclusion Criteria:

1. Current diagnosis of an additional neurologic condition such as Multiple Sclerosis, Parkinson disease, stroke, or brain injury
2. Severe illness or infection, including non-healing decubitus ulcers, untreated bladder or urinary tract infections, cardiovascular disease, lung disease, active heterotopic ossification, or uncontrolled hypertension
3. Severe neuropathic pain
4. Known pregnancy
5. Severe recurrent autonomic dysreflexia

Exclusion for involvement in TMS - History of seizure disorder, uncontrolled migraines, presence of cardiac pacemaker, metal implants in skull, medications that lower seizure threshold.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in motor evoked potential | Baseline, and 45-60 minutes after intervention on AIH day, AIHH day, and Sham AIH day
  The change in peak-to-peak amplitude of the motor evoked potential of the diaphragm will be tested using transcranial magnetic stimulation.
Change in maximal inspiratory pressure | Baseline, 1 day, 3 days, and 7 days after intervention blocks (daily AIH + respiratory strength training, daily AIHH + respiratory strength training, daily sham AIH + respiratory strength training.)
  Maximal inspiratory pressure is a non-invasive measure of the maximal force achieved when breathing in against an occluded airway.
Change in maximal expiratory pressure | Baseline, 1 day, 3 days, and 7 days after intervention blocks (daily AIH + respiratory strength training, daily AIHH + respiratory strength training, daily sham AIH + respiratory strength training.)
  Maximal expiratory pressure is a non-invasive measure of the maximal force achieved when breathing out against an occluded airway.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Fox, DPT, MHS, PhD, Principal Investigator — University of Florida & Brooks Rehabilitation
Locations (1):
- Brooks Rehabilitation, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No